CLINICAL TRIAL: NCT00503828
Title: The Efficacy and Safety of Derris Scandens Benth Extract and Naproxen for Therapy of Patients With Knee Osteoarthritis
Brief Title: Derris Scandens Benth Extract VS Naproxen in Knee OA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Ministry of Health, Thailand (Other Government)
Responsible Party: Department of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Siriraj CEU 50-001
Record Dates: First submitted 2007-07-18; First posted 2007-07-19 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2009-06

CONDITIONS: Knee Osteoarthritis
Keywords: Derris Scandens Benth extract; Osteoarthritis; WOMAC; 6-minute walk
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis | interventions — Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- naproxen (Active Comparator): Naproxen 500 mg/day for 4 weeks
  Interventions: Drug: naproxen
- Derris Scandens Benth (Experimental): Derris Scandens Benth
  Interventions: Drug: Derris scandens Benth extracts

INTERVENTIONS:
Drug: Derris scandens Benth extracts — Derris scandens Benth extracts (oral) 400 mg twice per day for 4 weeks
  Arms: Derris Scandens Benth
Drug: naproxen — Naproxen 500 mg/day for 4 weeks
  Arms: naproxen

SUMMARY:
Derris Scandens Benth (family : Leguminosae) is a woody vine growing throughout Southeast Asia, including Thailand. The stem of D.Scandens has been widely use in Thai traditional medicine, foe example of myalgia. Previous study shown that D.Scandens Benth extract has the anti-inflammatory activity. Although NSAIDs are efficaciously in the treatment of osteoarthritis,but the GI side effect is still concerned. In this study we aim to investigate the efficacy and safety of D. Scandens Benth extract compared with Naproxen for therapy of patients with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age >=50 yr
* Known case of primary knee osteoarthritis
* WOMAC pain subscale (item1) >= 5
* signed informed consent

Exclusion Criteria:

* hypersensitive to NSAIDs
* history of peptic ulcer or melena
* unable to walk , i.e. patient with severe spinal stenosis, myocardial infarction
* history of intra-articular injection of knee within 3 months
* status post knee replacement

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
WOMAC score | 2, 4 weeks

SECONDARY OUTCOMES:
6-minute walk, Quality of Life, adverse event | 2, 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Vilai Kuptniratsaikul, Assoc.Prof., Principal Investigator — Department of Rehabilitation Medicine, Faculty of Medicine Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkoknoi, Bangkok, Thailand